CLINICAL TRIAL: NCT03716310
Title: Impaired Platelet Reactivity as an Early Biomarker for Sepsis-related Thrombocytopenia
Brief Title: Platelet Reactivity in Septic Shock
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, MD, Università degli Studi di Ferrara
Other Study IDs: Sepsisplt
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Septic Shock; Thrombocytopenia; Sepsis; Platelet Aggregation; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Shock, Septic; Thrombocytopenia; Sepsis; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- septic shock patients: Inclusion criteria of the study were diagnosis of septic shock and a platelet count >150*103/mcL.
  Interventions: Diagnostic Test: platelet responsiveness evaluation

INTERVENTIONS:
Diagnostic Test: platelet responsiveness evaluation — Blood samples were anticoagulated with 0.129 mmol/L of sodium citrate and then centrifugated for 10 min at 200 rpm; platelets aggregation was assessed with an AggRAM Advanced Modular System light transmittance aggregometer (Helena Laboratories, Beaumont, Texas, USA). Low-molecular-weight heparin (LMWH) was given at least 8 hours before any blood aggregation sample. Agonist used to initiate aggregation test were: -Adenosine diphosphate (ADP) to assess P2Y12-dependent platelet aggregation; (20 ng) - Arachidonic acid (AA) to assess cyclooxygenase-dependent platelet Adenosine diphosphate aggregation (1 mcg) - thrombin receptor-activating peptide-6 (TRAP-6) to assess protease-activated receptor 1-dependent platelet aggregation. Max aggregation reached (Aggmax), the slope of the curve (slope) and the latency time (lat) were analyzed for each agonist.

SUMMARY:
Coagulation disorders and thrombocytopenia are common in patients with septic shock. Despite the clinical relevance of sepsis-induced thrombocytopenia, few studies have focused on the prediction of thrombocytopenia in this setting. The aim of this study was to evaluate whether platelets aggregometry and markers of platelets activation, such as mean platelet volume or platelet volume distribution width, could predict sepsis-induced thrombocytopenia in patients with septic shock and normal platelet count on the day of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of septic shock
* platelet count >150*103/mcL.

Exclusion Criteria:

* age <18 years
* history of any hematologic disorder
* chronic liver failure
* previous chemotherapy
* transfusion of platelet during the previous 4 weeks
* renal replacement therapy before ICU admission
* history of antiplatelet therapy during the 8 days before inclusion
* history of heparin-induced thrombocytopenia (HIT) or other acquired or induced thrombocytopenia
* occurrence of HIT (defined as HIT score over 3)
* active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care unit
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Occurence of sepsis-induced thrombocytopenia | 5 days after study inclusion
  Occurence of platelet count <150 *103/μL

SECONDARY OUTCOMES:
life-threatening bleeding | After 28 days from study inclusion
90-day mortality | after 90 days from study enrollment
number of Red blood cells (RBC) packs transfused during ICU stay | After 28 days from study inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Campo G, Valgimigli M, Gemmati D, Percoco G, Tognazzo S, Cicchitelli G, Catozzi L, Malagutti P, Anselmi M, Vassanelli C, Scapoli G, Ferrari R. Value of platelet reactivity in predicting response to treatment and clinical outcome in patients undergoing primary coronary intervention: insights into the STRATEGY Study. J Am Coll Cardiol. 2006 Dec 5;48(11):2178-85. doi: 10.1016/j.jacc.2005.12.085. Epub 2006 Nov 13. PMID 17161242
- [Background] Dewitte A, Lepreux S, Villeneuve J, Rigothier C, Combe C, Ouattara A, Ripoche J. Blood platelets and sepsis pathophysiology: A new therapeutic prospect in critically [corrected] ill patients? Ann Intensive Care. 2017 Dec 1;7(1):115. doi: 10.1186/s13613-017-0337-7. PMID 29192366